CLINICAL TRIAL: NCT04077320
Title: Neurological Changes With a Memory Self-efficacy Training Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Western BrainsCAN (Unknown)
Responsible Party: Principal Investigator, Lindsay Nagamatsu, Assistant Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BSCAN1920
Record Dates: First submitted 2019-08-28; First posted 2019-09-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: memory; older adults; randomized control trial; MRI; memory education
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware of the content of alternate groups. Both arms will be described as "Learning and Aging" groups to the participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memory Self-Efficacy Training (Experimental): Memory self-efficacy group training classes.
  Interventions: Behavioral: Memory Self-Efficacy Training
- General Education Group (Active Comparator): General education group classes (e.g., exercise, diet, sustainability, tc.)
  Interventions: Behavioral: General Education

INTERVENTIONS:
Behavioral: Memory Self-Efficacy Training — The intervention will consist of a six-week cognitive behavioral intervention integrating the four pillars of self-efficacy, Mastery, Social Modeling, Coaching, and Physiological Responses (West et al. 2008). Each week will comprise of a 1.5 hour session which focuses on an educational component, discussions and active learning practice activities to apply lesson material. Additionally, participants will be given take home exercises to practice outside a classroom setting. The sessions will be conducted in small groups of 4-6 people.
  Arms: Memory Self-Efficacy Training
Behavioral: General Education — The active control intervention will be a general education class consisting of real world knowledge and factual information on various topics unrelated to memory. This intervention will follow the same format as the memory self-efficacy training arm. One 1.5 hours session every week for 6 weeks, in small groups.
  Arms: General Education Group

SUMMARY:
Confidence in one's ability to accomplish a task, more formally known as self-efficacy, is an important psychological variable that can influence how the investigators perform on various tasks. Previous studies have shown that self-efficacy is a modifiable trait that can be improved and bolstered with training and practice. More importantly for this study, memory self-efficacy has been shown to be modifiable for older adults, consequently improving their performance on memory tasks. While there is evidence to support the importance of memory self-efficacy for successful memory performance in older adults, the underlying neurological changes that accompany these performance changes have not been explored. The goal of this study is to examine the changes in brain activity before and after a memory self-efficacy training program to better understand the mechanisms of both memory and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjective memory complaints within past 5 years
2. Objective memory impairment below age norms on standardized cognitive testing
3. Score below 25 on Montreal Cognitive Assessment
4. Scores 1.5 standard deviations below age norms on memory testing
5. Unimpaired performance in Activities of Daily Living
6. Intact general cognition
7. Fluently read, write and speak English
8. Right handed

Exclusion Criteria:

1. Co-morbidity that would impact cognition (depression, anxiety, stroke)
2. Prior diagnosis of dementia of any type
3. Use of prescription or recreational drug use that would impact cognition (excluding hormone replacement therapy)
4. Uncorrected visual or auditory deficits/impairments
5. Current participation in alternate study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Neurological bio-markers: Regional activation | Pre and Post intervention - 6 weeks
  Using fMRI identify changes in activation patterns or signal change when performing an associative memory task
Neurological bio-markers: Default mode network | Pre and Post intervention - 6 weeks
  Using fMRI during a resting state observe changes in default mode network activation

SECONDARY OUTCOMES:
Story Recall - Trained memory performance task | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were specifically practiced in the training intervention. Recall of a short story to estimate episodic memory capacity.
List Recall - Trained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were specifically practiced in the training intervention. Recall of a visually presented list of unrelated words to estimate episodic memory capacity and working memory.
Face-Name Pairs - Trained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were specifically practiced in the training intervention. Recall of a face-name pairs to evaluate associative memory.
RAVLT - Untrained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were not specifically practiced in the training intervention.
  Participants are asked to recall a list of verbally presented words immediately after presentation and after a delay. Used to evaluate sort term verbal memory and long term memory
Visual Spatial Learning Task - Untrained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were not specifically practiced in the training intervention.
  Subjects are given time to learn the location and design of shapes on a 6 x 4 matrix. Subjects are required to correctly select the 7 correct shapes from a selection of 15 and place them on the grid. Used to measure visual spatial memory
Digit Span Task - Untrained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were not specifically practiced in the training intervention.
  A series of numbers are verbally presented, increasing in length for the participant to repeat back. Measures working memory
Face-Scene Pairs - Untrained memory performance tasks | Pre and Post intervention - 6 weeks
  Observe the changes in memory performance using measures that were not specifically practiced in the training intervention.
  An alternative form of evaluating associative memory ability. Participants will be given face and scene pairs to remember.

OTHER OUTCOMES:
Memory self-efficacy: Multifactorial Memory Questionnaire (MMQ) | Pre and Post intervention - 6 weeks
  Multifactorial Memory Questionnaire (MMQ), 5-point scale Likert questions (min 0, max 4) evaluating subjective memory satisfaction, ability and strategy use.
  Satisfaction: 18 questions. Raw scores can be converted to T Scores using the normative data presented in MMQ administration and scoring manual. Converted T-Scores can range from 15 to 85. T-scores between 40-60 are considered normal relative to the population. While those below 40 are considered low scores and those above 60 high scores.
  Ability: 20 questions. Raw scores can be converted to T Scores using the normative data presented in MMQ administration and scoring manual. Interpretation of T-scores same as above sub-scale.
  Strategy: 19 questions. Raw scores can be converted to T Scores using the normative data presented in MMQ administration and scoring manual. Interpretation of T-scores same as above sub-scale.
  Each of the three MMQ scales is scored and interpreted separately.
Memory self-efficacy: Memory Self-efficacy Questionnaire (MSEQ) subjective scale | Pre and Post intervention - 6 weeks
  Memory self efficacy will be evaluated and compared between groups to evaluate the efficacy of each intervention arm. As there is no one measure that is the gold standard for memory self-efficacy two validated measures will be used for comparison.
  Measure by 2) Memory Self-efficacy Questionnaire (MSEQ) subjective scale of participant's confidence in completing various memory related tasks.
  Each task is scored by percent confidence of successfully completing the task (0 - 100%) Total memory self-efficacy is calculated by summing each task and taking the average. Values closer to 0% represent a worse overall memory self-efficacy, while values closer to 100% represent better memory self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Community, London, Ontario, Canada